CLINICAL TRIAL: NCT07090291
Title: China Colorectal Cancer Screening Trial 1 (C-Cost1): Colonoscopy Versus FIT Versus FIT Plus Blood Test in the Average Risk Population
Brief Title: China Colorectal Cancer Screening Trial 1 (C-Cost1)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Ding Ke-Feng, Professor, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: C-Cost1
Record Dates: First submitted 2025-07-20; First posted 2025-07-29 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer; Advanced Adenoma
Keywords: FIT; FIT plus blood test; cfDNA methylation; Colorectal cancer; Advanced colorectal adenoma; Early screening; Average risk population
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy; Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Colonoscopy group (Active Comparator): The internationally recommended screening protocol is adopted. The participants will only undergo a colonoscopy once at the first year. Suspicious lesions detected during the colonoscopy will be resected and further sent for pathological examination. All the participants will then receive annual follow-ups for the next 3 years, followed by long-term follow-ups.
  Interventions: Diagnostic Test: Colonoscopy
- FIT group (Active Comparator): The internationally recommended screening protocol is adopted. In the first 4 years of the screening phase, all participants will receive annual FIT tests. Participants with positive FIT results are recommended to undergo diagnostic colonoscopy. Suspicious lesions detected during the colonoscopy will be resected and further sent for pathological examination. Participants who refuse FIT tests, have negative FIT tests, have positive FIT tests but do not receive diagnostic colonoscopy will be screened again in the first 4 years. All the participants will be followed by long-term follow-ups.
  Interventions: Diagnostic Test: FIT
- FIT plus blood test group (Experimental): A new screening protocol is adopted. In the first 4 years of the screening phase, all participants will receive annual FIT tests and blood tests. Participants with positive FIT tests or positive blood tests are recommended to undergo diagnostic colonoscopy. Suspicious lesions detected during the colonoscopy will be resected and further sent for pathological examination. Participants who refuse FIT plus blood tests, have negative FIT plus blood tests, have positive FIT tests or positive blood tests but do not receive diagnostic colonoscopy will be screened again in the first 4 years. All the participants will be followed by long-term follow-ups.
  Interventions: Diagnostic Test: FIT; Diagnostic Test: Blood test

INTERVENTIONS:
Diagnostic Test: Colonoscopy — Colonoscopy is used to examine the inner lining of the colon and rectum. During the procedure, if suspicious growths (e.g., polyps) are detected, they will be biopsied and sent for pathological examination.
  Arms: Colonoscopy group
Diagnostic Test: FIT — FIT stands for Fecal Immunochemical Test, a non-invasive screening tool used primarily to detect hidden blood in the stool, which may indicate colorectal cancer or precancerous polyps. Positive cut-off level: 100 ng/mL.
  Arms: FIT group; FIT plus blood test group
Diagnostic Test: Blood test — Blood test based on cfDNA methylation will be performed.
  Arms: FIT plus blood test group

SUMMARY:
Colorectal cancer (CRC) is one of the most common malignancies in China. Currently, its incidence rate is increasing at a rate of 4% per year, exceeding the global annual average growth rate. Screening and early diagnosis of colorectal cancer and precancerous lesions are key measures to reduce the disease burden of colorectal cancer in China. In previous clinical studies, colorectal cancer screening in high risk population received extensive attention. However, it cannot be ignored that the majority of sporadic colorectal cancers occur in the average risk population. Therefore, there is an urgent need to develop new approach for colorectal cancer screening in the average risk population in China.

Fecal Immunochemical Testing (FIT) initial screening followed by diagnostic colonoscopy is widely recommended by colorectal cancer screening guidelines worldwide. The current colorectal cancer screening approach faces challenges including limited sensitivity of initial screening technologies and insufficient population coverage in organized screening programs in China. As initial screening technologies, non-invasive blood tests which detects cfDNA methylation have been reported to have higher accuracy than FIT in detecting colorectal cancer. However, There is a lack of randomized controlled trials (RCTs) comparing the effectiveness of colonoscopy, FIT and FIT plus blood test for colorectal cancer screening.

In China Colorectal Cancer Screening Trial 1 (C-Cost1), we propose to perform a multicenter, cluster randomized, parallel group trial directly comparing colonoscopy with FIT and with FIT plus blood test in the average risk population in China. The main research hypotheses are: (1) The screening protocol of FIT group (Group B) is non-inferior to the colonoscopy group (Group A) in the colorectal cancer mortality rate at 10 years; (2) The screening protocol of FIT plus blood test group (Group C) is superior to the FIT group (Group B) in the colorectal cancer mortality rate at 10 years. Either of the two hypotheses being met is acceptable.

DETAILED DESCRIPTION:
This study intends to recruit participants who meet the above inclusion and exclusion criteria in China, with the goal of recruiting at least 62200 eligible participants at baseline. The study adopts a cluster randomized controlled design. After signing the informed consent form, eligible participants will be randomly assigned to 3 colorectal cancer screening groups. All participants will undergo a 4-year screening phase, and then all participants will be followed up for a long term. Fecal, blood, and tissue samples will be collected from the participants during the study. The grouping and specific intervention measures are as follows:

1. Colonoscopy group (n = 22600): The internationally recommended screening protocol is adopted. The participants will only undergo a colonoscopy once at the first year. Suspicious lesions detected during the colonoscopy will be resected and further sent for pathological examination. All the participants will then receive annual follow-ups for the next 3 years, followed by long-term follow-ups.
2. FIT group (n = 22600): The internationally recommended screening protocol is adopted. In the first 4 years of the screening phase, all participants will receive annual FIT tests. Participants with positive FIT results are recommended to undergo diagnostic colonoscopy. Suspicious lesions detected during the colonoscopy will be resected and further sent for pathological examination. Participants who refuse FIT tests, have negative FIT tests, have positive FIT tests but do not receive diagnostic colonoscopy will be screened again in the first 4 years. All the participants will be followed by long-term follow-ups.
3. FIT plus blood test group (n = 17000): A new screening protocol is adopted. In the first 4 years of the screening phase, all participants will receive annual FIT tests and blood tests. Participants with positive FIT tests or positive blood tests are recommended to undergo diagnostic colonoscopy. Suspicious lesions detected during the colonoscopy will be resected and further sent for pathological examination. Participants who refuse FIT plus blood tests, have negative FIT plus blood tests, have positive FIT tests or positive blood tests but do not receive diagnostic colonoscopy will be screened again in the first 4 years. All the participants will be followed by long-term follow-ups.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 45-74 years old;
2. In good general condition, with normal mental state and voluntarily signing the informed consent form;

Exclusion Criteria:

1. Personal history of colorectal cancer or precancerous lesions;
2. History of previous colonrectal resection surgery;
3. Diagnosed with cancer before enrollment or currently receiving any cancer-related treatment;
4. Having received colonoscopy, flexible sigmoidoscopy, CT colonography and other examinations within the past 5 years;
5. Having received FIT or FIT-sDNA or cfDNA test within the past 1 year;
6. Symptomatic lower gastrointestinal diseases or symptoms suggesting the need for diagnostic colonoscopy for confirmation;
7. Accompanied by severe diseases that are not suitable for colorectal cancer screening;

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62200 (Estimated)
Dates: Start 2025-08-08 (Actual); Primary Completion 2035-07 (Estimated); Study Completion 2035-07 (Estimated)

PRIMARY OUTCOMES:
Mortality rate of colorectal cancer | 10 years
  Mortality rate of colorectal cancer

SECONDARY OUTCOMES:
Detection rate of advanced colorectal neoplasms | 4 years
  Advanced colorectal neoplasms includes advanced adenomas and colorectal cancer
Population compliance rate | 4 years
  Population compliance rate
Proportion of colorectal cancer at different stages | 4 years
  Proportion of colorectal cancer at different stages
Incidence rate of colorectal cancer | 10 years
  Incidence rate of colorectal cancer
Quality of life (QOL) | 4 years
  Quality of life will be assessed by EuroQol five-dimensional questionnaire (EQ-5D）
Total cost and cost per detected lesion | 4 years
  Total cost and cost per detected lesion
Incremental cost-effectiveness ratio | 4 years
  Incremental cost-effectiveness ratio

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The Fourth Hospital of Hebei Medical University, Hebei
  - Nanjing Medical University, Nanjing

IPD SHARING:
Plan to Share IPD: No